CLINICAL TRIAL: NCT04501757
Title: Expanded Access Use of Naxitamab/GM-CSF Immunotherapy for Consolidation of Complete Remission or Relapsed/Refractory High-Risk Neuroblastoma
Brief Title: Naxitamab and GM-CSF in People With Neuroblastoma
Status: No longer available | Type: Expanded Access
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-227
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: High-Risk Neuroblastoma
Keywords: Remission High-Risk Neuroblastoma; Relapsed/Refractory High-Risk Neuroblastoma; Naxitamab; GM-CSF; 20-227
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Naxitamab/GM-CSF — naxitamab/GM-CSF for 5 Cycles

SUMMARY:
This is an Expanded Access Program (EAP) that will give the participants access to the drug naxitamab before it is approved by the FDA. Naxitamab will be combined with granulocyte-macrophage colony stimulating factor (GM-CSF). Participants in this study will have high-risk neuroblastoma that either went away completely after treatment (complete remission) or has come back (relapsed/refractory).

Researchers think the combination of naxitamab and GM-CSF will be effective because naxitamab and GM-CSF strengthen the immune system's response to cancer cells in different ways. Naxitamab is an antibody, like the proteins made by the immune system to protect the body from harm. Naxitamab helps the cells of the immune system to find and attack cancer cells. GM-CSF is a protein that strengthens the immune system by increasing the number of immune cells called granulocytes. Granulocytes are white blood cells that fight off cancer cells. The combination of naxitamab and GM-CSF is a type of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are ineligible to participate in study NCT03363373 (IRB# 18-375), will be considered for treatment under this expanded access protocol.
* Diagnosis of NB as defined by a) histopathology (confirmed by the MSK Department of Pathology), or b) BM metastases or MIBG-avid lesion(s) plus high urine catecholamine levels
* Patients must have HR-NB (MYCN-amplified stage 2/3/4/4S of any age and MYCNnonamplified stage 4 in patients greater than 18 months of age).
* Patients must be in first or greater CR or have refractory or relapsed disease
* If previously treated with any anti-GD2 mAb, human anti-hu3F8 antibody (HAHA) titer must be negative.

Exclusion Criteria:

* Active life-threatening infection
* Pregnant women or women who are breastfeeding
* HAHA titer positive
* History of anaphylaxis CTCAE grade 4 to naxitamab

Min Age: 18 Months | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm